CLINICAL TRIAL: NCT06495580
Title: Optimizing Visual Outcomes: Use of Optic Nerve Stimulation in Endoscopic Cranial Approaches
Brief Title: Optic Nerve Stimulation To Prevent Visual Deficits After Endoscopic Cranial Approaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-41739
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Optic Nerve Injuries; Sellar Tumor; Skull Base Neoplasms
MeSH Terms: conditions — Optic Nerve Injuries; Skull Base Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will enroll adult (18 y.o. and older) patients undergoing open or endonasal endoscopic surgery for suprasellar tumors including meningiomas, craniopharyngiomas and pituitary adenomas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optic Nerve Stimulation (Experimental): The most significant procedure will be using an anterograde microstimulator and provoke stimulations to the optic nerve as the surgery proceeds. During surgery, the optic nerve and chiasm will be stimulated and the response recorded in both eyes and occipital cortex via skin electrodes. These responses will be monitored at all times by the neuromonitorig team who will inform if changes in neural responses change. The use of microstimulator has been proven safe in other surgical approaches.
  Interventions: Procedure: Optic Nerve Stimulation
- No Intervention (No Intervention): Patients receiving regular standard of care in endoscopic endonasal approaches within the same case series.

INTERVENTIONS:
Procedure: Optic Nerve Stimulation — Anterograde Stimulation of the Optic Neve.
  Arms: Optic Nerve Stimulation

SUMMARY:
Assessing the function of the optic nerve is paramount during various neurosurgical procedures. Effective optic nerve monitoring has remained elusive as Visual Evoked Potentials (the current existing tool) provides only diffuse and delayed assessment of nerve function. Here, the investigators propose a prospective study involving adult patients (aged 18 years and older) undergoing endonasal or open cranial approaches around the optic nerves, who will receive pre- and post-operative visual evaluations. During surgery, the optic nerve and chiasm will be stimulated, and the response will be recorded in both eyes and the occipital cortex via skin electrodes. The investigators aim to utilize anterograde optic nerve microstimulation to assess the nerve's integrity during open and endoscopic cranial approaches. Electrophysiological readings will be acquired, as is routine in the operating room, by our team of experts, and intraoperative findings will be correlated with post- surgical clinical outcomes. Our objective is to utilize existing technology in the operating room to safely and effectively monitor optic nerve function during surgery.

DETAILED DESCRIPTION:
Our hypothesis is that utilizing anterograde optic nerve microstimulation during open and endoscopic cranial approaches will allow for more accurate and real-time assessment of optic nerve function compared to the current standard of Visual Evoked Potentials. The investigators predict that this novel approach will lead to improved intraoperative monitoring and better correlation with post- surgical clinical outcomes.

The study design proposed is interventional and prospective. It involves implementing a novel approach, anterograde optic nerve microstimulation, during surgical procedures to assess optic nerve integrity. This design entails actively intervening during the surgical process to stimulate the optic nerve and record responses, indicating an interventional approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with suprasellar tumors including meningiomas, craniopharyngiomas and pituitary adenomas.
* Must not present with any permanent or temporal visual deficit.
* Must receive an open or endoscopic endonasal procedure as part of their care.

Exclusion Criteria:

* Preexisting visual impairments unrelated to the tumor.
* History of prior cranial surgeries or radiation therapy.
* Significant cognitive impairment or inability to provide informed consent
* Contraindications to microstimulation procedures such as uncontrolled coagulopathy or active infection.
* Patients with tumors located outside the sellar region or those requiring emergent or urgent surgery due to life-threatening complications.
* Additionally, individuals with systemic conditions or comorbidities that may significantly impact visual function or surgical outcomes, such as uncontrolled diabetes mellitus or severe cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Visual Deficits | 6 weeks after surgery date.
  Patients that received our intervention will be evaluated post operatively for regular standard of care six weeks post-operatively. During visual evaluation, the PI of this study will determine post-operative visual field and visual acuity. These parameters will be compared to pre-operative visual acuity and visual field status.

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Goldschmidt, MD, PhD, Principal Investigator — UCSF Department of Neurological Surgery
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margalit NS, Lesser JB, Moche J, Sen C. Meningiomas involving the optic nerve: technical aspects and outcomes for a series of 50 patients. Neurosurgery. 2003 Sep;53(3):523-32; discussion 532-3. doi: 10.1227/01.neu.0000079506.75164.f4. PMID 12943569
- [Background] Cohen AR, Cooper PR, Kupersmith MJ, Flamm ES, Ransohoff J. Visual recovery after transsphenoidal removal of pituitary adenomas. Neurosurgery. 1985 Sep;17(3):446-52. doi: 10.1227/00006123-198509000-00008. PMID 4047355
- [Background] Jashek-Ahmed F, Cabrilo I, Bal J, Sanders B, Grieve J, Dorward NL, Marcus HJ. Intraoperative monitoring of visual evoked potentials in patients undergoing transsphenoidal surgery for pituitary adenoma: a systematic review. BMC Neurol. 2021 Jul 23;21(1):287. doi: 10.1186/s12883-021-02315-4. PMID 34301198
- [Background] Newman S. A prospective study of cavernous sinus surgery for meningiomas and resultant common ophthalmic complications (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2007;105:392-447. PMID 18427624
- [Background] Carnevale JA, Babu CS, Goldberg JL, Fong R, Schwartz TH. Visual deterioration after endonasal endoscopic skull base surgery: causes, treatments, and outcomes. J Neurosurg. 2021 Oct 1;136(4):1103-1113. doi: 10.3171/2021.3.JNS204378. Print 2022 Apr 1. PMID 34598134
- [Background] Sakata K, Komaki S, Takeshige N, Negoto T, Kikuchi J, Kajiwara S, Orito K, Nakamura H, Hirohata M, Morioka M. Visual Outcomes and Surgical Approach Selection Focusing on Active Optic Canal Decompression and Maximum Safe Resection for Suprasellar Meningiomas. Neurol Med Chir (Tokyo). 2023 Sep 15;63(9):381-392. doi: 10.2176/jns-nmc.2021-0142. Epub 2023 Jul 10. PMID 37423756
- [Background] Chung SB, Park CW, Seo DW, Kong DS, Park SK. Intraoperative visual evoked potential has no association with postoperative visual outcomes in transsphenoidal surgery. Acta Neurochir (Wien). 2012 Aug;154(8):1505-10. doi: 10.1007/s00701-012-1426-x. Epub 2012 Jun 29. PMID 22739773
- [Background] Qiao N, Yang X, Li C, Ma G, Kang J, Liu C, Cao L, Zhang Y, Gui S. The predictive value of intraoperative visual evoked potential for visual outcome after extended endoscopic endonasal surgery for adult craniopharyngioma. J Neurosurg. 2021 May 7;135(6):1714-1724. doi: 10.3171/2020.10.JNS202779. Print 2021 Dec 1. PMID 33962373
- [Background] Benedicic M, Bosnjak R. Intraoperative monitoring of the visual function using cortical potentials after electrical epidural stimulation of the optic nerve. Acta Neurochir (Wien). 2011 Oct;153(10):1919-27. doi: 10.1007/s00701-011-1098-y. Epub 2011 Aug 5. PMID 21818643
- [Background] Sasaki T, Itakura T, Suzuki K, Kasuya H, Munakata R, Muramatsu H, Ichikawa T, Sato T, Endo Y, Sakuma J, Matsumoto M. Intraoperative monitoring of visual evoked potential: introduction of a clinically useful method. J Neurosurg. 2010 Feb;112(2):273-84. doi: 10.3171/2008.9.JNS08451. PMID 19199497
- [Background] Benedicic M, Bosnjak R. Optic nerve potentials and cortical potentials after stimulation of the anterior visual pathway during neurosurgery. Doc Ophthalmol. 2011 Apr;122(2):115-25. doi: 10.1007/s10633-011-9265-2. Epub 2011 Mar 16. PMID 21409432